CLINICAL TRIAL: NCT01886339
Title: SNIF (Sniff Nasal Inspiratory Force) REFERENCE VALUES OF MEDITERRANEAN POPULATION.
Acronym: SNIF REF V
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: 09/117/1031
Record Dates: First submitted 2013-06-21; First posted 2013-06-25 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Healthy People Programs

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy population
  Interventions: Other: SNIF test (Sniff Nasal Inspiratory Force)

INTERVENTIONS:
Other: SNIF test (Sniff Nasal Inspiratory Force)

SUMMARY:
SNIF test has been described as a method to explore the diaphragmatic function. But there are no defined the reference values of this test in healthy population. The investigators' hypothesis is that there is a variation on SNIF values in Mediterranean population depending on gender, age and anthropometric variables such as height and weight.

The investigators will analyze 1000 SNIF test of healthy people. The investigators will divide in 5 groups of age (20-30, 30-40, 40-50, 50-60, 60-70) and in each group the investigators will study 100 men and 100 women.

All the subjects will perform a forced spirometry, maximal inspiratory pressure (MIP) and SNIF. If spirometry and MIP are correct the investigators will consider that person has a correct diaphragmatic function and strength. Then the investigators will measure the SNIF test. With all of these SNIF values the investigators will try to achieve the reference values of this test in the different groups of age in Mediterranean population. And the investigators will compare SNIF with MIP.

Cross multicentric study. Hospitals involved: Hospital de Bellvitge, Hospital del Mar, Hospital Parc Taulí, Hospital de la Santa Creu i Sant Pau (coordinator center) and Hospital de la Vall d'Hebrón.

ELIGIBILITY:
Inclusion Criteria:

* Healthy people with spirometry and MIP values in the reference range
* Age between 20 and 70 years old
* Caucasian race

Exclusion Criteria:

* Rhinitis
* Nasal obstruction
* Frequent episodes of epistaxis
* Ongoing cold

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 439 (Actual)
Dates: Start 2010-06; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
SNIF test | Basal
  Main objectives:
  * To define the SNIF reference values in a healthy Mediterranean population.
  * Analyze the influence of different variables such as gender, age, height and weight on this measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided